CLINICAL TRIAL: NCT01160952
Title: Long-term Versus Short-term Sequential Therapy (Intravenous Itraconazole Followed by Oral Solution) of Itraconazole as Primary Prophylaxis in Patients Undergoing Allogeneic Stem Cell Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Renmin Hospital of Zhongshan Guangdong (Unknown); Zhujiang Hospital (Other)
Responsible Party: Jian Liu (President of the hospital), Guangzhou General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPO-I-08-CN-041-C; ITRFUN4046 (Other Grant/Funding Number: Xi'an Janssen pharmaceutical Ltd.)
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2010-07

CONDITIONS: Hematological Diseases; Allogeneic Stem Cell Transplantation
Keywords: primary prophylaxis; itraconazole; stem cell transplantation
MeSH Terms: conditions — Hematologic Diseases | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- long-term group (Other): long-term group refers to prophylaxis by using itraconazole for up to 90 days
  Interventions: Drug: itraconazole
- short term group (Other): short term group refers to prophylaxis by itraconazole for 30 days
  Interventions: Drug: itraconazole

INTERVENTIONS:
Drug: itraconazole — the two groups are defined by different treatment duration

SUMMARY:
* The primary objective of this study is to evaluate the efficacy and safety profile of itraconazole as in primary prophylaxis
* The second objective of this study is to find the difference between long-term versus short-term sequential therapy of Itraconazole (intravenous followed by oral itraconazole) as primary prophylaxis of invasive fungal infections (IFI) in patients undergoing allogeneic stem cell transplantation (allo-SCT)
* also to explore the relationship between the incidence of IFI with plasma concentrations of itraconazole and hydroxy-itraconazole

DETAILED DESCRIPTION:
Invasive fungal infections (IFI) remain the major cause of death among neutropenic patients receiving high dose chemotherapy or allo-SCT. Especially, patients undergoing allo-SCT generally receive intensive immunosuppressive therapy, which make those patients at high risk of developing IFI.

Prompt intensive antifungal therapy may increase the incidence rate of IFI and improved responses and survival. Antifungal prophylaxis has been recommended in patients undergoing allo-SCT by Infectious diseases society of America (IDSA) and Chinese guidelines for the diagnosis and management of IFI in patients with hematologic/malignant tumor (revised).

Few studies have addressed the role of previous IFI in the feasibility of stem cell transplant, or the secondary prophylaxis with antifungal drugs in preventing recurrence of infection after transplantation. However, given the lack of prospective studies, the role of primary antifungal prevention and the course of treatment remain unclear.

Itraconazole is a wide-spectrum triazole antifungal agent active against Candida albicans, non-albicans, Aspergillus spp., Blastomyces dermatitidis, Blastomyces coccidioides, Cryptococcus neoformans, Sporothrix schenkii, Paracoccidioides brasiliensis, Histoplasma spp. and various kinds of yeast fungi and mycetes.

The role of itraconazole in IFI prophylaxis has been proved by many interventional studies. However the optimal course of prophylaxis is still unknown，especially in China. In this prospective, multicentric study of primary antifungal prevention, long-term or short-term sequential therapy (intravenous followed by oral itraconazole) will be given at standard dose to patients undergoing allogeneic stem cell transplantation to assess the efficacy and safety of itraconazole in primary prophylaxis, and to analysis the relationship between the incidence rate of IFI with plasma concentrations of itraconazole and hydroxy-itraconazole.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between 14 and 60 years of age, inclusive
* Patients who affected by hematological diseases, receiving allo-SCT
* Patients with no previous proven or probable invasive fungal infections. Patients without microbiological evidence but with effective anti-fungal therapy history are inclusive
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Currently taking the contra-indicated medications such as teldane, astemizol, cisapride and HMG-CoA reductase inhibitor（e.g. Simvastatin, lovastatin, oral Midazolam and Triazolam）
* History of allergy or intolerance to imidazole or azoles anti-fungal agents (e.g. Fluconazol, Itraconazole, Ketoconazole, Miconazole, Clotrimazole)
* Pregnant women, lactating women or women of child bearing potential without applying valid contraceptive measures
* Patients with current cardiac dysfunction (especially with congestive heart failure) or with the history of congestive heart failure
* Patients with severe liver dysfunction (aminotransferase levels >= 5 times the upper limit of normal and total bilirubin level >= 3mg/dL(51.3 μmol/L); or the severity of liver dysfunction does not match this criteria but the patient is in bad condition and not suitable for this trial( doctors make the decision);
* Patients with renal insufficiency having serum Ccr level <30ml/min, calculated from the following formula:

Male: Ccr (ml/min)=(140-age)×weight (kg) /(0.8136×Crea (μmol/L) ) Female:Ccr (ml/min)=(140-age)×weight (kg) ×0.85/(0.8136× Crea (μmol/L) )

* Patients received any experimental drug within 14 days before the planned start of treatment.
* Patients with bad whole body status and not suitable for the trial (doctors make the decision)

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-12 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
efficacy evaluation | 90 days
  the success rate of prophylaxis therapy by itraconazole

SECONDARY OUTCOMES:
group difference evaluation | 90 days
  efficacy difference between long-term and short-term groups per success rate at day 90

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xiao, MD, Principal Investigator — Guangzhou General Hospital of Guangzhou Military Command
Locations (1):
- Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Marr KA, Crippa F, Leisenring W, Hoyle M, Boeckh M, Balajee SA, Nichols WG, Musher B, Corey L. Itraconazole versus fluconazole for prevention of fungal infections in patients receiving allogeneic stem cell transplants. Blood. 2004 Feb 15;103(4):1527-33. doi: 10.1182/blood-2003-08-2644. Epub 2003 Oct 2. PMID 14525770
- [Background] Winston DJ, Maziarz RT, Chandrasekar PH, Lazarus HM, Goldman M, Blumer JL, Leitz GJ, Territo MC. Intravenous and oral itraconazole versus intravenous and oral fluconazole for long-term antifungal prophylaxis in allogeneic hematopoietic stem-cell transplant recipients. A multicenter, randomized trial. Ann Intern Med. 2003 May 6;138(9):705-13. doi: 10.7326/0003-4819-138-9-200305060-00006. PMID 12729424
- [Background] Chinese guideline for the diagnosis and management of IFI in patients with hematologic/maliglant tumor (revised). Chinese journal of internal medicine 2007，46(7):607-610.
- [Derived] Lin R, Xu X, Li Y, Sun J, Fan Z, Jiang Q, Huang F, Zhou H, Nie D, Guo Z, Mao Y, Xiao Y, Liu Q. Comparison of long-term and short-term administration of itraconazole for primary antifungal prophylaxis in recipients of allogeneic hematopoietic stem cell transplantation: a multicenter, randomized, open-label trial. Transpl Infect Dis. 2014 Apr;16(2):286-94. doi: 10.1111/tid.12192. Epub 2014 Mar 5. PMID 24593273